CLINICAL TRIAL: NCT01470430
Title: Study to Measure Systemic VEGF Levels in ROP Infants Following Intravitreal Anti-VEGF Therapy or Retinal Laser Treatment
Brief Title: VEGF In Systemic Circulation Of ROP-infants
Status: Withdrawn | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Andreas Stahl, MD, MD, University Hospital Freiburg
Other Study IDs: VISOR Study
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ROP infants treated with intravitreal anti-VEGF agents
- ROP infants treated with retinal laser photocoagulation

SUMMARY:
The purpose of this study is to measure systemic levels of vascular endothelial growth factor (VEGF) and other proteins (e.g. IGF-1) in the systemic circulation of infants with retinopathy of prematurity (ROP) following ocular treatment with either intravitreal injections of anti-VEGF agents or retinal laser photocoagulation. The primary aim is to determine if serum VEGF levels change after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of retinopathy of prematurity requiring treatment

Exclusion Criteria:

* Anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: prematurely born infants with retinopathy of prematurity requiring treatment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Systemic VEGF levels following treatment | 16 weeks
  comparing VEGF levels in serum of ROP infants treated with intravitreal anti-VEGF agents vs. retinal laser photocoagulation over 16 weeks post treatment

SECONDARY OUTCOMES:
Systemic levels of other growth factors (e.g. IGF-1) | 16 weeks
  comparing systemic levels of other (non-VEGF) factors in serum of ROP infants treated with intravitreal anti-VEGF agents vs. retinal laser photocoagulation

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Stahl, MD, Principal Investigator — University Eye Hospital Freiburg, Germany
Locations (1):
- University Eye Hospital, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- See also: University Eye Hospital Freiburg, Germany — http://www.uniklinik-freiburg.de/augenklinik/live/homede.html?weiterleitung=ja